CLINICAL TRIAL: NCT07268560
Title: Aztreonam-Avibactam Real World Study Against Metallo-β-lactamase-Producing Carbapenem-Resistant Enterobacterales
Brief Title: Real-World Effectiveness of Aztreonam-Avibactam Against MBL-Producing CRE
Acronym: AWARE
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 98628137
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Complicated Intra-Abdominal Infections, cIAIs; Hospital-acquired Pneumonia (HAP); Ventilator-Associated Pneumonia (VAP)
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized adult patients with MBL-producing CRE infections treated with ATM-AVI.: The study population consists of hospitalized adult patients with MBL-producing CRE infections treated with ATM-AVI. Investigators will start eligibility screening and recruitment from adult patients who have received ≥24 hours of ATM-AVI.
  Interventions: Drug: Aztreonam-Avibactam

INTERVENTIONS:
Drug: Aztreonam-Avibactam — Hospitalized adult patients with MBL-producing CRE infections treated with ATM-AVI.

SUMMARY:
Why This Study is Needed Some bacterial infections have become resistant to common antibiotics, making them very difficult to treat. This is a growing and serious health problem. A new combination drug, Aztreonam-Avibactam (we'll call it ATM-AVI), has been developed to fight these tough bacteria.

This new drug was recently approved for use in Europe (April 2024), the United States (February 2025), and China (June 2025). Because it is so new, there is very little information available, especially in China, on how well it works for real patients outside of initial testing.

This lack of real-world experience means we don't know enough about:

* How effective it is for typical patients in China.
* The types of patients and infections it is used for.
* How it affects a patient's time in the hospital. This study aims to fill these gaps by looking at how ATM-AVI performs in Chinese hospitals, which will help doctors better treat these dangerous infections and improve patient recovery.

What the Study Aims to Find Out

Main Goal:

To see how well ATM-AVI works for adult patients in China with these specific antibiotic-resistant infections.

Other Goals:

To gather more details about:

* How patients are responding to the treatment at different points (e.g., after 5 days, at the end of treatment, and at a follow-up check).
* Whether the bacteria causing the infection are cleared.
* How the treatment affects the patient's hospital stay and use of resources.
* The number of patients who, unfortunately, pass away during or after treatment.
* The characteristics of the patients (like age) and their infections.
* How doctors are using this new drug and if it's used alongside other antibiotics.

How the Study Will Work This is an observational study that will be conducted in about 30 hospitals across China. We plan to include around 100 adult patients who were hospitalized with these tough infections and received the new drug, ATM-AVI, for at least one full day.

The study will run from October 2025 to June 2027. We will look at both past (retrospective) and future (prospective) patients. For past patients, we will review their existing medical records. For future patients, we will ask for their permission (informed consent) before collecting any information.

We will collect information from patient records, such as:

* Basic patient details and the nature of their infection.
* How and when the ATM-AVI drug was used.
* Details about their hospital stay.
* The results of their lab tests. A doctor will assess and record how each patient is doing at key points: 5 days after starting the drug, at the end of the treatment, and at a follow-up check to see if the infection is cured.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 years or older 2. Hospitalized with a diagnosis of confirmed cIAI or HAP/VAP 3. Confirmed infection with MBL-producing CRE 4. Received on label use of ATM-AVI treatment for ≥24 hours 5. Informed consent will be obtained or waived.

Exclusion Criteria:

* 1. Confirmed or suspected infection caused by Gram-negative species not expected to respond to ATM-AVI 2. Currently enrolled in an interventional clinical tria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of hospitalized adult patients with MBL-producing CRE infections treated with ATM-AVI. Investigators will start eligibility screening and recruitment from adult patients who have received ≥24 hours of ATM-AVI.
  The index date is defined as the ATM-AVI initiation date, for which the date of first administration is used. The baseline period spans from 14 days before the index date to the index date, or from the date of admission to the index date, whichever is later. The observations will be both retrospective and prospective. Patients will be followed from ATM-AVI use until death, study withdrawal, or hospital discharge, whichever occurs first. For patients discharged before Day 28, a phone follow-up is necessary for assessment of the 28-day all-cause mortality.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy outcome measure is the proportion of patients who had a clinical response of clinical success, failure, and indeterminate, respectively, which will be assessed at the EOT visit. | From enrollment to the end of treatment at 4 weeks
  The primary descriptive efficacy analysis will be the estimate of the clinical response rate along with nominal 95% CIs using the Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The study will include interim report and a final clinical study report. Upon completion of the study and finalization of the study report, the results of this NI study will be submitted for publication and/or posted in a publicly accessible results database. Publications will adhere to the recommendations of the International Committee of Medical Journal Editors (ICMJE).